CLINICAL TRIAL: NCT02831907
Title: Assessment of Portal Flow Using Bedside Doppler Ultrasonography for the Detection of Portal Pulsatility as a Risk Factor for Acute Kidney Injury in Cardiac Surgery Patients
Brief Title: Portal Flow Pulsatility as a Risk Factor for Acute Kidney Injury After Cardiac Surgery
Acronym: PP-AKI
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Principal Investigator, Andre Denault, MD PhD FRCPC ABIM-CCM, Montreal Heart Institute
Other Study IDs: 2016-1946
Record Dates: First submitted 2016-07-05; First posted 2016-07-13 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: C.Surgical Procedure; Cardiac; Acute Kidney Injury; Postoperative Complications; Right-Sided Heart Failure; Cardio-Renal Syndrome
Keywords: Ultrasonography; Portal vein Doppler; Renal Doppler; Cardio-Intestinal syndrome; Delirium; Renal congestion; Intra-renal hemodynamics
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications; Heart Failure; Cardio-Renal Syndrome; Delirium | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: Adult patients having a cardiac surgery at the Montreal Heart Institute
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — All cardiac surgery procedures with the use of cardiopulmonary bypass

SUMMARY:
The purpose of this study is to evaluate the possible association between portal vein flow pulsatility and acute kidney injury after cardiac surgery. Participants will undergo assessment of portal vein flow and intra-renal blood flow using bedside Doppler ultrasound before surgery and daily for three days after cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury is a frequent complication after cardiac surgery. Venous congestion from right ventricular dysfunction and fluid overload can impair kidney perfusion resulting in the cardio-renal syndrome.

An increase in the variation of blood flow velocity in the portal vein during the cardiac cycle called portal pulsatility is a sign of congestive heart failure. Portal pulsatility occurs when increased central venous pressure results liver venous congestion. The presence of abnormal portal pulsatility could be used as a marker of venous congestions in other organs such as the kidneys. Discontinuous intra-renal vein flow is a risk factor for death or re-hospitalization in heart failure patients and could be seen in patients with portal pulsatility.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Undergoing cardiac surgery with the use of cardiopulmonary bypass
* Able to provide consent.

Exclusion Criteria:

* Chronic renal replacement therapy before the procedure.
* Chronic kidney disease stage 5 defined as a estimated glomerular filtration rate by the MDRD equation (eGFR-MDRD) of 15 mL/min/1,73m2 or less.
* Critical pre-operative state defined as aborted sudden death, preoperative cardiac massage, preoperative ventilation before anaesthetic room, preoperative inotropes or intra-aortic counterpulsation balloon.
* Patients previously diagnosed with a condition interfering with Doppler evaluation of the portal system: Portal vein thrombosis, Cirrhosis.
* Patients with documented AKI before surgery.
* Confirmed or suspected pregnancy.
* Kidney transplant recipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective or urgent cardiac surgery with the use of cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury defined by an increase in serum creatinine of ≥150% of baseline or an elevation of 0.3 mg/dL or more within a contiguous period of 48 hours. (KDIGO criteria) | 7 days after surgery
  The definition of acute kidney injury is based on the KDIGO guidelines

SECONDARY OUTCOMES:
Mortality | 30 days after surgery
Duration of intensive care stay | 30 days after surgery
Delirium defined as an Intensive Care Delirium Screening Checklist score of 4 or more. | 7 days after surgery
  Intensive Care Delirium Screening Checklist is a validated tool for the screening of delirium in the intensive care unit.
Composite endpoint of persistent organ dysfunction (POD) plus death at day 3 and 7 | 3 days and 7 days after surgery
  Persistent organ dysfunction (POD) plus death is a validated outcome measure in cardiac surgery patients. It is defined as one of the following: mechanical ventilation without breaks for a period of more than 48 hours or vasopressor therapy (ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin, dopamine 45 μg/ kg/min, or phenylephrine 450 μg/min for more than 2 hours in a given day); or mechanical circulatory support (ongoing need for mechanical devices such as extracorporeal membrane oxygenation or intra-aortic counterpulsation balloon pump) or continuous renal replacement therapy or new intermittent hemodialysis; or death.
Severe acute kidney injury (KDIGO stage 2 or more) defined by an increase in serum creatinine of ≥200% of baseline. | 7 days after surgery
  The definition of acute kidney injury is based on the KDIGO guidelines
Discontinuous blow flow in renal interlobar vessels | 3 days after surgery
  The presence of abnormal discontinuous blow flow in renal interlobar vessels assessed by bedside Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: André Denault, MD, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prowle JR, Echeverri JE, Ligabo EV, Ronco C, Bellomo R. Fluid balance and acute kidney injury. Nat Rev Nephrol. 2010 Feb;6(2):107-15. doi: 10.1038/nrneph.2009.213. Epub 2009 Dec 22. PMID 20027192
- [Background] McNaughton DA, Abu-Yousef MM. Doppler US of the liver made simple. Radiographics. 2011 Jan-Feb;31(1):161-88. doi: 10.1148/rg.311105093. PMID 21257940
- [Background] Catalano D, Caruso G, DiFazzio S, Carpinteri G, Scalisi N, Trovato GM. Portal vein pulsatility ratio and heart failure. J Clin Ultrasound. 1998 Jan;26(1):27-31. doi: 10.1002/(sici)1097-0096(199801)26:13.0.co;2-l. PMID 9475205
- [Background] Bouchard J, Soroko SB, Chertow GM, Himmelfarb J, Ikizler TA, Paganini EP, Mehta RL; Program to Improve Care in Acute Renal Disease (PICARD) Study Group. Fluid accumulation, survival and recovery of kidney function in critically ill patients with acute kidney injury. Kidney Int. 2009 Aug;76(4):422-7. doi: 10.1038/ki.2009.159. Epub 2009 May 13. PMID 19436332
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Taylor DO, Starling RC, Young JB, Tang WHW. Importance of venous congestion for worsening of renal function in advanced decompensated heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):589-596. doi: 10.1016/j.jacc.2008.05.068. PMID 19215833
- [Background] Styczynski G, Milewska A, Marczewska M, Sobieraj P, Sobczynska M, Dabrowski M, Kuch-Wocial A, Szmigielski C. Echocardiographic Correlates of Abnormal Liver Tests in Patients with Exacerbation of Chronic Heart Failure. J Am Soc Echocardiogr. 2016 Feb;29(2):132-9. doi: 10.1016/j.echo.2015.09.012. Epub 2015 Nov 6. PMID 26549056
- [Background] Iida N, Seo Y, Sai S, Machino-Ohtsuka T, Yamamoto M, Ishizu T, Kawakami Y, Aonuma K. Clinical Implications of Intrarenal Hemodynamic Evaluation by Doppler Ultrasonography in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):674-82. doi: 10.1016/j.jchf.2016.03.016. Epub 2016 May 11. PMID 27179835
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney inter., Suppl. 2012; 2: 1-138.
- [Background] Heyland DK, Muscedere J, Drover J, Jiang X, Day AG; Canadian Critical Care Trials Group. Persistent organ dysfunction plus death: a novel, composite outcome measure for critical care trials. Crit Care. 2011;15(2):R98. doi: 10.1186/cc10110. Epub 2011 Mar 18. PMID 21418560
- [Background] Stoppe C, McDonald B, Benstoem C, Elke G, Meybohm P, Whitlock R, Fremes S, Fowler R, Lamarche Y, Jiang X, Day AG, Heyland DK. Evaluation of Persistent Organ Dysfunction Plus Death As a Novel Composite Outcome in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):30-8. doi: 10.1053/j.jvca.2015.07.035. Epub 2015 Jul 29. PMID 26847748
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542